CLINICAL TRIAL: NCT03898492
Title: Quality Assessment of a Training Period for Physical and Mentally Disabled People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOU-UU-2018-001
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Disabled Persons; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: One intervention group and one control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The participants in this group participated in exercise two times/week for 8 weeks
  Interventions: Other: Physical training
- Control (No Intervention): The participants in the control group were instructed to maintain their daily routines.

INTERVENTIONS:
Other: Physical training — Training two times/week for an hour each time in 8 weeks. The training included strength training, aerobic training, balance training and flexibility training. The training was modified to the participants and initiated by the staff at the center.
  Arms: Intervention

SUMMARY:
The aim of the study was to evaluate the effect of a 8 week training period compared with control group in physical and mentally disabled adults. The effect was evaluated in relation to their physical status. Furthermore, physical activity was measured using steps and active minutes.

DETAILED DESCRIPTION:
This study aimed at making a quality assessment of a 8 week training period for adults with physical and mental disabilities. A control group was added to compare the effect of the training with no training. Before the training period the participants were tested in relation to their physical status: weight, height, fat%, blood pressure, Aastrand test, chair stand test and waist circumference. In addition to this, the participants were instructed to wear an accelerometer to measure step and active minutes for 2-3 days a work.

The staff at the day center, where the participants works in daytime, were responsible for the physical training 2 times/week for 8 weeks. The training was an hour of combined aerobic, strength, balance and flexibility training.

The participants were tested after the training period using the same test-protocol as before.

ELIGIBILITY:
Inclusion Criteria:

* User of the centers included in the study
* Being able to stand alone
* Being able to use an exercise bike
* Being able to understand danish

Exclusion Criteria:

* Pregnancy
* Pacemaker
* Not being able to stand up by themselves

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Body mass index | Through study completion, an average of 8 weeks
  weight (kg)/height (m) x height (m)
Blood pressure | Through study completion, an average of 8 weeks
  Diastolic pressure (mmHg) Systolic pressure (mmHg)
Completed chair stands | Through study completion, an average of 8 weeks
  Number of completed chair stands
Aastrand test | Through study completion, an average of 8 weeks
  Bike test to measure the physical fitness.
Waist circumference | Through study completion, an average of 8 weeks
  Measured in cm
Physical activity | During test session - 2-3 days
  Number of steps and active minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Drachmann, Msc, Study Director — University College of Northern Jutland, Denmark. Department of Physiotherapy
Locations (1):
- Department of Physiotherapy, University College of Northern Jutland, Aalborg, Denmark